CLINICAL TRIAL: NCT00004993
Title: Can PTH Reverse Glucocorticoid-induced Osteoporosis
Brief Title: Can Parathyroid Hormone Injections Reverse Glucocorticoid-induced Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: LANENE (completed); DK46661
Record Dates: First submitted 2000-03-17; First posted 2000-03-20 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Osteoporosis
Keywords: Parathyroid hormone (1-34); Glucocorticoid-induced osteoporosis; Postmenopausal women; osteoporotic fractures
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures | interventions — Parathyroid Hormone; Teriparatide

INTERVENTIONS:
Drug: Parathyroid hormone (hPTH 1-34)

SUMMARY:
Glucocorticoids are potent anti-inflammatory and immunosuppressive agents. However, prolonged use of these potent agents results in severe bone loss and osteoporotic fractures. Parathyroid hormone (1-34), when given as a daily injection has been found to dramatically increase bone mass in osteoporotic animals and postmenopausal women. The purpose of this study is to determine whether 2 years of daily PTH (1-34) injections will increase bone mass and reduce the development of new fractures. In addition, we will follow the study subjects for 2 more years to determine which type of anti-resorptive agent is required to maintain the newly formed bone.

We are enrolling postmenopausal women that are on chronic corticosteroid therapy (prednisone etc.) and have bone loss (osteopenia by DXA) to be a part of this four-year-long study. The patients will receive two-year therapy with either PTH (1-34) or placebo, and for the second part of the study subjects receive either estrogen and placebo or alendronate and placebo. We will measure bone gain by standard bone densitometry, special x-rays of the spine and hip, and serum and urine bone markers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women on glucocorticoids (prednisone 5mg/d or greater
* Osteopenia by T score of hip or lumbar spine of -2.0
* All study subjects must be on a stable dose of estrogen/progesterone or raloxifene
* Ambulatory and able to come to the clinical center 9 times over 2 years
* Willing to sign an informed consent

Exclusion Criteria:

* Generalized disease of the bone (other than glucocorticoid-induced osteoporosis), including hyperparathyroidism, hyperthyroidism, Paget's disease)
* Diseases that affect bone metabolism (e.g. alcoholism, inflammatory bowel disease, malabsorption, renal disease (Cr2) or liver disease (transaminase level 2 times limit of normal)
* Within the past 1 year, regular use of medications that are known to affect bone metabolism (e.g. anabolic steroids, anticoagulants, anticonvulsants, pharmacologic doses of vitamin D and vitamin A supplements).
* History of drug abuse
* Senile dementia, paraplegia and/or quadriplegia
* Unstable rheumatic disease with clinically significant renal or central nervous system involvement.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08; Study Completion 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: Qaiser Rehman, M.D., Study Director — University of California at San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Lane NE, Sanchez S, Modin GW, Genant HK, Pierini E, Arnaud CD. Parathyroid hormone treatment can reverse corticosteroid-induced osteoporosis. Results of a randomized controlled clinical trial. J Clin Invest. 1998 Oct 15;102(8):1627-33. doi: 10.1172/JCI3914. PMID 9788977